CLINICAL TRIAL: NCT01218438
Title: A Clinical Study of Immune Globulin Subcutaneous (Human), 20% Solution (IGSC, 20%) for the Evaluation of Efficacy, Safety, Tolerability and Pharmacokinetics in Subjects With Primary Immunodeficiency Diseases (PIDD)
Brief Title: Phase 2/3 Study of IGSC, 20% in PIDD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170904
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Results first posted 2017-02-15 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Primary Immunodeficiency Diseases (PID)
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — gamma-Globulins; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Epochs 1-4 (Experimental): Epoch 1 (13 weeks): Pharmacokinetic (PK) assessment at 2nd to last infusion (in all participants ≥12 years of age). Participants will be treated intravenously once every 3 or 4 weeks at same monthly equivalent dose as prior to the study.
  Epoch 2 (12-16 weeks): PK assessment (in first 15 participants ≥12 years of age) at 9th infusion to determine adjusted dose for Epoch 3 and individually adapted dose for Epoch 4. Participants will be treated subcutaneously every 7 days at a dose of IGSC, 20% that is 145% of the weekly equivalent of the IV dose in Epoch 1.
  Epoch 3 (12 weeks): Participants will be treated subcutaneously every 7 days using the adjusted dose determined in Epoch 2. The individually adapted dose for use in Epoch 4 will also be determined.
  Epoch 4 (40 weeks): Participants will be treated subcutaneously once every week at the individually adapted dose determined in Epoch 3. PK assessment at 17th infusion.
  Interventions: Biological: Immune Globulin Intravenous (Human), 10% Solution; Drug: Immune Globulin Subcutaneous (Human), 20% Solution

INTERVENTIONS:
Biological: Immune Globulin Intravenous (Human), 10% Solution — Intravenous infusion with IGIV, 10%
  Other Names: IGIV; 10%
Drug: Immune Globulin Subcutaneous (Human), 20% Solution — Subcutaneous infusion with IGSC, 20%
  Other Names: IGSC; 20%

SUMMARY:
The purpose of this study is to develop a 20% subcutaneous (SC) immunoglobulin preparation for the treatment of patients with primary immunodeficiency diseases (PIDD).

ELIGIBILITY:
Main Inclusion Criteria:

* Documented diagnosis of a form of primary humoral immunodeficiency involving defective antibody formation and requiring gammaglobulin replacement as defined according to the IUIS Scientific Committee, 2011 and by diagnostic criteria according to Conley et al. (1999). The diagnosis must be confirmed by the Medical Director prior to first treatment with the investigational product (IP) in the study.
* Participant is 2 years or older at the time of screening, and has a minimum body weight of 13 kg.
* Written informed consent has been obtained from either the participant or the participant's legally authorized representative prior to any study-related procedures and study product administration
* Participant has been receiving a stable monthly equivalent dose of IgG at an average minimum dose equivalent to 300 mg/kg bodyweight (BW)/4 weeks and a maximum dose equivalent to 1.0 gram/kg BW/4 weeks, for a minimum of 12 weeks prior to first treatment with the IP in the study.
* Serum trough level of IgG > 500 mg/dL at screening
* Participant is willing and able to comply with the requirements of the protocol

Main Exclusion Criteria:

* Participant has known history of or is positive at screening for one or more of the following: hepatitis B surface antigen (HBsAg), polymerase chain reaction (PCR) for Hepatitis C virus(HCV), PCR for human immunodeficiency virus (HIV) Type 1/2
* Abnormal laboratory values at screening meeting any one of the following criteria (abnormal tests may be repeated once to determine if they are persistent):

  * Persistent alanine aminotransferase (ALT) and aspartate amino transferase(AST) > 2.5 times the upper limit of normal for the testing laboratory
  * Persistent severe neutropenia (defined as an absolute neutrophil count [ANC] ≤500/mm^3)
* Creatinine clearance (CLcr) value that is < 60% of normal for age and gender either measured, or calculated according to the Cockcroft-Gault formula
* Malignancy (other than adequately treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix), unless the disease-free period prior to screening exceeds 5 years
* Participant is receiving anti-coagulation therapy (low dose aspirin at ≤325 mg/day is permitted) or has a history of thrombotic episodes (including deep vein thrombosis, myocardial infarction, cerebrovascular accident, pulmonary embolism) or sickle cell disease with crisis within 12 months prior to screening or a history of thrombophilia
* Abnormal protein loss (protein losing enteropathy, nephrotic syndrome)
* Anemia that would preclude phlebotomy for laboratory studies according to standard practice at the site
* Acute serious bacterial infection within 3 months prior to screening
* Ongoing history of hypersensitivity or persistent reactions (urticaria, breathing difficulty, severe hypotension, or anaphylaxis) following intravenous immunoglobulin, subcutaneous immunoglobulin, and/or Immune Serum Globulin (ISG) infusions
* Severe immunoglobulin A (IgA) deficiency (less than 0.07g/L) with known anti-IgA antibodies and a history of hypersensitivity
* Participant is on continuous systemic antibacterial antibiotics at doses sufficient to treat or prevent bacterial infections, and, in the opinion of the investigator, cannot stop these for the duration of the study without putting the patient at risk of increased infections
* Participant has active infection and is receiving antibiotic therapy for the treatment of infection at the time of screening
* Bleeding disorder or thrombocytopenia with a platelet count less than 20,000/μL, or who, in the opinion of the investigator, would be at significant risk of increased bleeding or bruising as a result of subcutaneous therapy
* Total protein > 9 g/dL or myeloma or macroglobulinemia (IgM) or paraproteinemia
* Severe dermatitis that would preclude adequate sites for safe product administration
* Women of childbearing potential meeting any one of the following criteria:

  * Participant presents with a positive pregnancy test
  * Participant is breast feeding
  * Participant intends to begin nursing during the course of the study
  * Participant does not agree to employ adequate birth-control measures (e.g. intrauterine device, diaphragm or condom [for male partner] with spermicidal jelly or foam, or birth control pills/patches) throughout the course of the study
* Participation in another clinical study and exposure to an investigational product or device within 30 days prior to study enrollment (exception: treatment in a previous Baxter immunoglobulin study)
* Participant is scheduled to participate in another (non-Baxter) non-observational (interventional) clinical study involving an investigational product or device during the course of the study

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2013-01-28 (Actual); Primary Completion 2015-03-13 (Actual); Study Completion 2015-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (18):
- United States (16):
  - University of California, Irvine, Irvine, California
  - IMMUNOe International Research Centers, Centennial, Colorado
  - Allergy Associates of the Palm Beaches, North Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Family Allergy and Asthma Research Institute, Louisville, Kentucky
  - Children's Hospital New Orleans- LSUHSC School of Medicine, New Orleans, Louisiana
  - Midwest Immunology Clinical and Infusion Center, Plymouth, Minnesota
  - SSM Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Montefiore Medical Center Division of Allergy/Immunology, The Bronx, New York
  - Oklahoma Institute of Allergy and Asthma Clinical Research, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - Dallas Allergy Immunology Research, Dallas, Texas
  - Allergy Asthma and Immunology Clinic PA, Irving, Texas
  - Rocky Mountain Asthma/Allergy/Immunology, Layton, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Centre Hospitalier Universitaire (CHU) Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital- McGill University health Center, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Background] Al-Herz W, Bousfiha A, Casanova JL, Chapel H, Conley ME, Cunningham-Rundles C, Etzioni A, Fischer A, Franco JL, Geha RS, Hammarstrom L, Nonoyama S, Notarangelo LD, Ochs HD, Puck JM, Roifman CM, Seger R, Tang ML. Primary immunodeficiency diseases: an update on the classification from the international union of immunological societies expert committee for primary immunodeficiency. Front Immunol. 2011 Nov 8;2:54. doi: 10.3389/fimmu.2011.00054. eCollection 2011. PMID 22566844
- [Background] Conley ME, Notarangelo LD, Etzioni A. Diagnostic criteria for primary immunodeficiencies. Representing PAGID (Pan-American Group for Immunodeficiency) and ESID (European Society for Immunodeficiencies). Clin Immunol. 1999 Dec;93(3):190-7. doi: 10.1006/clim.1999.4799. No abstract available. PMID 10600329
- [Derived] Li Z, McCoy B, Engl W, Yel L. Steady-State Serum IgG Trough Levels Are Adequate for Pharmacokinetic Assessment in Patients with Immunodeficiencies Receiving Subcutaneous Immune Globulin. J Clin Immunol. 2021 Aug;41(6):1331-1338. doi: 10.1007/s10875-021-00990-z. Epub 2021 May 26. PMID 34036490
- [Derived] Suez D, Krivan G, Jolles S, Stein M, Gupta S, Paris K, van Hagen PM, Brodszki N, Engl W, Leibl H, McCoy B, Yel L. Safety and tolerability of subcutaneous immunoglobulin 20% in primary immunodeficiency diseases from two continents. Immunotherapy. 2019 Aug;11(12):1057-1065. doi: 10.2217/imt-2019-0057. Epub 2019 Jul 3. PMID 31268374
- [Derived] Gupta S, Stein M, Hussain I, Paris K, Engl W, McCoy B, Rabbat CJ, Yel L. Tolerability of Ig20Gly during onboarding in patients with primary immunodeficiency diseases. Ann Allergy Asthma Immunol. 2019 Sep;123(3):271-279.e1. doi: 10.1016/j.anai.2019.06.004. Epub 2019 Jun 20. PMID 31228628
- [Derived] Paris K, Haddad E, Borte M, Brodszki N, Derfalvi B, Marodi L, Hussain I, Darter A, Engl W, Leibl H, McCoy B, Yel L. Tolerability of subcutaneous immunoglobulin 20%, Ig20Gly, in pediatric patients with primary immunodeficiencies. Immunotherapy. 2019 Apr;11(5):397-406. doi: 10.2217/imt-2018-0088. Epub 2019 Jan 9. PMID 30626238
- [Derived] Suez D, Stein M, Gupta S, Hussain I, Melamed I, Paris K, Darter A, Bourgeois C, Fritsch S, Leibl H, McCoy B, Gelmont D, Yel L. Efficacy, Safety, and Pharmacokinetics of a Novel Human Immune Globulin Subcutaneous, 20 % in Patients with Primary Immunodeficiency Diseases in North America. J Clin Immunol. 2016 Oct;36(7):700-12. doi: 10.1007/s10875-016-0327-9. Epub 2016 Aug 31. PMID 27582171

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled (signed informed consent) at 15 sites.
Pre-assignment Details: A total of 86 participants provided informed consent. 9 of these participants did not start Epoch1, of which there were 6 screen failures; 2 were not able to receive their first infusion according to protocol timeline; and 1 withdrew. Therefore, 77 participants started Epoch 1 of the study.
Groups:
- Study Participants: - EPOCH 1: (13 weeks): Pharmacokinetics (PK) at 2nd to last infusion (participants ≥12 years of age). Participants will be treated with immune globulin administered intravenously (IGIV), 10% once every 3 or 4 weeks at same monthly equivalent dose as prior to study. - EPOCH 2: (12-16 weeks): PK (first 15 participants ≥12 years of age) at 9th infusion to determine adjusted dose for Epoch 3 and individually adapted dose for Epoch 4. Participants will be treated with immune globulin administered subcutaneously (IGSC), 20% every 7 days at dose of IGSC, 20% that is 145% of the weekly equivalent of the IV dose in Epoch 1. - EPOCH 3: (12 weeks): Participants will be treated subcutaneously every 7 days using the adjusted dose determined in Epoch 2. The individually adapted dose for use in Epoch 4 will also be determined. - EPOCH 4: (40 weeks): Participants will be treated subcutaneously once every week at the individually adapted dose determined in Epoch 3. PK assessment at 17th infusion.
Period: Epoch 1
Arm/Group | Study Participants
Started | 77
Completed | 74
Not Completed | 3
Not completed — Physician Decision | 2
Not completed — Adverse Event | 1
Period: Epoch 2
Arm/Group | Study Participants
Started | 45
Completed | 45
Not Completed | 0
Period: Epoch 3
Arm/Group | Study Participants
Started | 74
Completed | 70
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 1
Period: Epoch 4
Arm/Group | Study Participants
Started | 70
Completed | 67
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Dataset: All participants who received at least one dose of immunoglobulin.
Groups:
- Study Epochs 1-4: - EPOCH 1: (13 weeks): Pharmacokinetics (PK) at 2nd to last infusion (participants ≥12 years of age). Participants will be treated with immune globulin administered intravenously (IGIV), 10% once every 3 or 4 weeks at same monthly equivalent dose as prior to study. - EPOCH 2: (12-16 weeks): PK (first 15 participants ≥12 years of age) at 9th infusion to determine adjusted dose for Epoch 3 and individually adapted dose for Epoch 4. Participants will be treated with immune globulin administered subcutaneously (IGSC), 20% every 7 days at dose of IGSC, 20% that is 145% of the weekly equivalent of the IV dose in Epoch 1. - EPOCH 3: (12 weeks): Participants will be treated subcutaneously every 7 days using the adjusted dose determined in Epoch 2. The individually adapted dose for use in Epoch 4 will also be determined. - EPOCH 4: (40 weeks): Participants will be treated subcutaneously once every week at the individually adapted dose determined in Epoch 3. PK assessment at 17th infusion.
Arm/Group | Study Epochs 1-4
Number analyzed (Participants) | 77
Age, Continuous [Median (Full Range); unit: Years] | 36.0 [3 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Rate of Acute Serious Bacterial Infections Per Year (ASBI)
Description: Annual rate of validated acute serious bacterial infections was calculated using a Poisson model to account for the different lengths of observation per participant. The observation period for each participant starts with the day of the first subcutaneous (SC) infusion in Study Epoch 2 and ends with the day of the End of Study visit.
Time Frame: 1 year
Population: Safety Analysis Set
Measure: Number; unit: Estimated infections/ year
Arm/Group | Study Participants
Number analyzed (Participants) | 74
Estimated infections/ year | 0.012
Statistical Analysis 1: Comparison: Study Participants; Test type: Superiority or Other; p < 0.0001, Poisson; Poisson = 0.012, 99% CI 1-sided [upper limit 0.024]

2. Secondary Outcome: Annual Rate of All Infections Per Participant
Time Frame: 1 year
Population: Safety Analysis Set
Measure: Number (95% Confidence Interval); unit: Estimated infections/year
Groups:
- Intravenous 10% - Epoch 1: - EPOCH 1: (13 weeks): Pharmacokinetics (PK) at 2nd to last infusion (participants ≥12 years of age). Participants will be treated with immune globulin administered intravenously (IGIV), 10% once every 3 or 4 weeks at same monthly equivalent dose as prior to study.
- Subcutaneous 20% - Epochs 2 Thru 4: - EPOCH 2: (12-16 weeks): PK (first 15 participants ≥12 years of age) at 9th infusion to determine adjusted dose for Epoch 3 and individually adapted dose for Epoch 4. Participants will be treated with immune globulin administered subcutaneously (IGSC), 20% every 7 days at dose of IGSC, 20% that is 145% of the weekly equivalent of the IV dose in Epoch 1. - EPOCH 3: (12 weeks): Participants will be treated subcutaneously every 7 days using the adjusted dose determined in Epoch 2. The individually adapted dose for use in Epoch 4 will also be determined. - EPOCH 4: (40 weeks): Participants will be treated subcutaneously once every week at the individually adapted dose determined in Epoch 3. PK assessment at 17th infusion.
Arm/Group | Intravenous 10% - Epoch 1 | Subcutaneous 20% - Epochs 2 Thru 4
Number analyzed (Participants) | 77 | 74
Estimated infections/year | 3.86 [2.77 to 5.22] | 2.41 [1.89 to 3.03]

3. Secondary Outcome: Annual Rate of Sinus Infections Per Participant
Time Frame: 1 year
Population: Safety Analysis Set
Measure: Number (99% Confidence Interval); unit: Estimated infections/year
Arm/Group | Intravenous 10% - Epoch 1 | Subcutaneous 20% - Epochs 2 Thru 4
Number analyzed (Participants) | 77 | 74
Estimated infections/year | 0.97 [0.61 to 1.45] | 0.69 [0.50 to 0.93]

4. Secondary Outcome: Annual Rate of Fever Episodes Per Participant
Time Frame: 1 year
Population: Safety Analysis Set
Measure: Number (95% Confidence Interval); unit: Estimated episodes/year
Arm/Group | Intravenous 10% - Epoch 1 | Subcutaneous 20% - Epochs 2 Thru 4
Number analyzed (Participants) | 77 | 74
Estimated episodes/year | 0.61 [0.34 to 0.99] | 0.13 [0.08 to 0.21]

5. Secondary Outcome: Annual Rate of Days Off School/Work or Days Unable to Perform Normal Daily Activities Due to Illness or Infection Per Participant
Time Frame: 1 year
Population: Safety Analysis Set
Measure: Number (95% Confidence Interval); unit: Estimated days off/participant
Arm/Group | Intravenous 10% - Epoch 1 | Subcutaneous 20% - Epochs 2 Thru 4
Number analyzed (Participants) | 77 | 74
Estimated days off/participant | 3.20 [1.88 to 5.03] | 1.16 [0.70 to 1.79]

6. Secondary Outcome: Annual Rate of Days on Antibiotics Per Participant
Time Frame: 1 year
Population: Safety Analysis Set
Measure: Number (95% Confidence Interval); unit: Estimated days/particpant
Arm/Group | Intravenous 10% - Epoch 1 | Subcutaneous 20% - Epochs 2 Thru 4
Number analyzed (Participants) | 77 | 74
Estimated days/particpant | 63.20 [43.39 to 88.29] | 57.59 [40.71 to 78.59]

7. Secondary Outcome: Annual Rate of Hospitalizations for Illness or Infection Per Participant
Time Frame: 1 year
Population: Safety Analysis Set
Measure: Number (95% Confidence Interval); unit: Estimated hospitalizations/participant
Arm/Group | Intravenous 10% - Epoch 1 | Subcutaneous 20% - Epochs 2 Thru 4
Number analyzed (Participants) | 77 | 74
Estimated hospitalizations/participant | 0.05 [0.02 to 0.10] | 0.02 [0.01 to 0.04]

8. Secondary Outcome: Annual Rate of Days of Hospitalizations for Illness or Infection Per Participant
Time Frame: 1 year
Population: Safety Analysis Set
Measure: Number (95% Confidence Interval); unit: Estimated days/participant
Groups:
- Intravenous 10% - Epoch 1: Epoch 1 (13 weeks): Pharmacokinetic (PK) assessment at 2nd to last infusion (in all participants ≥12 years of age). Participants will be treated intravenously once every 3 or 4 weeks at same monthly equivalent dose as prior to the study.
- Subcutaneous 20% - Epochs 2 Thru 4: Epoch 2 (12-16 weeks): PK assessment (in first 15 participants ≥12 years of age) at 9th infusion to determine adjusted dose for Epoch 3 and individually adapted dose for Epoch 4. Participants will be treated subcutaneously every 7 days at a dose of IGSC, 20% that is 145% of the weekly equivalent of the IV dose in Epoch 1. Epoch 3 (12 weeks): Participants will be treated subcutaneously every 7 days using the adjusted dose determined in Epoch 2. The individually adapted dose for use in Epoch 4 will also be determined. Epoch 4 (40 weeks): Participants will be treated subcutaneously once every week at the individually adapted dose determined in Epoch 3. PK assessment at 17th infusion.
Arm/Group | Intravenous 10% - Epoch 1 | Subcutaneous 20% - Epochs 2 Thru 4
Number analyzed (Participants) | 77 | 74
Estimated days/participant | 0.20 [0.08 to 0.42] | 0.11 [0.05 to 0.20]

9. Secondary Outcome: Annual Rate of Acute (Urgent or Unscheduled) Physician Visits, or Visits to the Emergency Room for Illness or Infection Per Participant
Time Frame: 1 year
Population: Safety Analysis Set
Measure: Number (95% Confidence Interval); unit: Estimated visits/participant
Arm/Group | Intravenous 10% - Epoch 1 | Subcutaneous 20% - Epochs 2 Thru 4
Number analyzed (Participants) | 77 | 74
Estimated visits/participant | 1.73 [1.03 to 2.68] | 0.86 [0.54 to 1.28]

10. Secondary Outcome: Bioavailability of IGSC, 20% as Measured by the Ratio of the Geometric Means of Immunoglobulin G (IgG) AUCSC (Epoch 4) to IgG AUCIV,0-τ (Standardized to 1 Week) (Epoch 1) Adjusted for Dose and Dosing Frequency (Participants ≥12 Years Old)
Description: IGSC, 20% = Immune Globulin Subcutaneous (Human), 20% Solution; AUCSC = area under the concentration-time curve following subcutaneous administration; AUCIV,0-τ = area under the concentration-time curve following intravenous administration over a dosing interval
Time Frame: Epoch 1: 3 week IV administration interval: Week 10, 11, 12, 13. Epoch 1: 4 week IV interval: Week 9, 10, 11, 12, 13. Epoch 4 Subcutaneous administration weeks 17, 18
Population: Safety Analysis Set with correctly administered IGIV 10% dose in Epoch 1
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Study Epochs 1-4
Number analyzed (Participants) | 49
Ratio | 1.0855 [1.0394 to 1.1336]

11. Secondary Outcome: Trough Levels of IgG (Total), and IgG Subclasses at the End of the Treatment Intervals
Time Frame: Epoch 1: 3 week IV interval- weeks 0, 1, 4, 7, 10, 13. Epoch 1: 4 week IV interval- weeks 0, 1, 5, 9, 13. Epochs 2 & 3: Subcutaneous (SC) weeks 5, 9. Epoch 4: SC weeks 1, 9, 17, 29, 40 (week dependent on time to establish "Adjusted Dose" in Epoch 2)
Population: Safety Analysis Set - sub-groups with data at relevant time points
Measure: Geometric Mean (95% Confidence Interval); unit: g/L
Groups:
- IV 10% 3 Weeks: Epoch 1 (13 weeks): Pharmacokinetic (PK) assessment at 2nd to last infusion (in all participants ≥12 years of age). Participants will be treated intravenously once every 3 or 4 weeks at same monthly equivalent dose as prior to the study. Epoch 2 (12-16 weeks): PK assessment (in first 15 participants ≥12 years of age) at 9th infusion to determine adjusted dose for Epoch 3 and individually adapted dose for Epoch 4. Participants will be treated subcutaneously every 7 days at a dose of IGSC, 20% that is 145% of the weekly equivalent of the IV dose in Epoch 1. Epoch 3 (12 weeks): Participants will be treated subcutaneously every 7 days using the adjusted dose determined in Epoch 2. The individually adapted dose for use in Epoch 4 will also be determined. Epoch 4 (40 weeks): Participants will be treated subcutaneously once every week at the individually adapted dose determined in Epoch 3. PK assessment at 17th infusion.
Arm/Group | IV 10% 3 Weeks | IV 10% 4 Weeks | SC 20% 145% IV 1 Week | SC 20% Adjusted 1 Week | SC 20% Individualized 1 Week
Number analyzed (Participants) | 19 | 50 | 27 | 66 | 57
g/L
  Total IgG | 11.58 [10.36 to 12.94] | 10.19 [9.55 to 10.88] | 14.77 [13.86 to 15.74] | 14.20 [13.48 to 14.96] | 14.74 [14.03 to 15.48]
  IgG Subclass 1 | 6.23 [5.47 to 7.09] | 5.45 [5.04 to 5.91] | 8.06 [7.51 to 8.65] | 7.83 [7.33 to 8.38] | 7.41 [6.98 to 7.87]
  IgG Subclass 2 | 3.92 [3.53 to 4.35] | 3.30 [3.08 to 3.54] | 4.83 [4.47 to 5.21] | 4.95 [4.65 to 5.26] | 4.94 [4.69 to 5.20]
  IgG Subclass 3 | 0.352 [0.285 to 0.435] | 0.405 [0.347 to 0.473] | 0.516 [0.463 to 0.574] | 0.514 [0.458 to 0.578] | 0.514 [0.456 to 0.580]
  IgG Subclass 4 | 0.239 [0.202 to 0.281] | 0.186 [0.165 to 0.209] | 0.309 [0.273 to 0.350] | 0.304 [0.280 to 0.331] | 0.311 [0.289 to 0.335]

12. Secondary Outcome: Trough Levels of Anti-Tetanus Antibody
Time Frame: Epoch 1: 3 week IV interval- weeks 1, 4, 7, 10, 13. Epoch 1: 4 week IV interval- weeks 1, 5, 9, 13. Epochs 2 & 3: Subcutaneous (SC) weeks 5, 9. Epoch 4: SC weeks 1, 9, 17, 29, 40 (week dependent on time to establish "Adjusted Dose" in Epoch 2)
Population: Safety Analysis Set - sub-groups with data at relevant time points
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 64
IU/mL
  Pre-Study Medication- Epoch 1 Week 1 (N= 64) | 2.28 [1.84 to 2.82]
  IV 10% 3 Weeks- Epoch 1 Week 4 (N= 15) | 3.36 [2.44 to 4.63]
  IV 10% 3 Weeks- Epoch 1 Week 7 (N= 16) | 2.66 [2.04 to 3.48]
  IV 10% 3 Weeks - Epoch 1 Week 10 (N= 19) | 2.55 [1.83 to 3.56]
  IV 10% 3 Weeks- Epoch 1 Week 13 (N= 16) | 2.26 [1.52 to 3.37]
  IV 10% 4 Weeks- Epoch 1 Week 5 (N= 46) | 1.92 [1.44 to 2.56]
  IV 10% 4 Weeks- Epoch 1 Week 9 (N= 44) | 2.31 [1.79 to 2.96]
  IV 10% 4 Weeks- Epoch 1 Week 13 (N= 43) | 2.28 [1.84 to 2.81]
  SC 20% 145% IV 1 Week- Epoch 2 Week 5 (N= 29) | 4.08 [3.12 to 5.33]
  SC 20% 145% IV 1 Week- Epoch 2 Week 9 (N= 27) | 4.49 [3.32 to 6.08]
  SC 20% adjusted 1 Week- Epoch 3 Week 5 (N= 55) | 3.76 [3.21 to 4.40]
  SC 20% adjusted 1 Week- Epoch 3 Week 9 (N= 58) | 3.09 [2.64 to 3.62]
  SC 20% adjusted 1 Week- Epoch 4 Week 1 (N= 62) | 2.75 [2.39 to 3.17]
  SC 20% individualized 1 Week Epoch 4 Week 9 (N=58) | 3.15 [2.73 to 3.63]
  SC 20% individualized 1 Week Epoch 4 Week 17(N=51) | 3.17 [2.74 to 3.67]
  SC 20% individualized 1 Week Epoch 4 Week 29(N=54) | 1.74 [1.48 to 2.03]
  SC 20% individualized 1 Week- End of Study (N= 53) | 1.97 [1.66 to 2.32]

13. Secondary Outcome: Trough Levels of Anti-Haemophilus Influenza B Antibody
Time Frame: as for outcome 12
Population: Safety Analysis Set - sub-groups with data at relevant time points
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 65
mg/L
  Pre-Study Medication- Epoch 1 Week 1 (N= 65) | 2.91 [2.55 to 3.34]
  IV 10% 3 Weeks- Epoch 1 Week 4 (N= 15) | 2.71 [2.07 to 3.56]
  IV 10% 3 Weeks- Epoch 1 Week 7 (N= 16) | 3.08 [2.36 to 4.01]
  IV 10% 3 Weeks- Epoch 1 Week 10 (N= 19) | 2.42 [1.75 to 3.36]
  IV 10% 3 Weeks- Epoch 1 Week 13 (N= 14) | 2.47 [1.85 to 3.29]
  IV 10% 4 Weeks- Epoch 1 Week 5 (N= 45) | 2.82 [2.30 to 3.46]
  IV 10% 4 Weeks- Epoch 1 Week 9 (N= 44) | 2.71 [2.23 to 3.30]
  IV 10% 4 Weeks- Epoch 1 Week 13 (N= 43) | 2.74 [2.20 to 3.42]
  SC 20% 145% IV 1 Week- Epoch 2 Week 5 (N= 29) | 4.07 [3.44 to 4.83]
  SC 20% 145% IV 1 Week- Epoch 2 Week 9 (N= 27) | 3.94 [3.30 to 4.71]
  SC 20% adjusted 1 Week- Epoch 3 Week 5 (N= 56) | 3.59 [3.12 to 4.14]
  SC 20% adjusted 1 Week- Epoch 3 Week 9 (N= 58) | 3.62 [3.10 to 4.22]
  SC 20% adjusted 1 Week- Epoch 4 Week 1 (N= 62) | 3.47 [3.06 to 3.94]
  SC 20% individualized 1 Week Epoch 4 Week 9 (N=58) | 4.35 [3.87 to 4.89]
  SC 20% individualized 1 Week Epoch 4 Week 17(N=51) | 4.76 [4.21 to 5.39]
  SC 20% individualized 1 Week Epoch 4 Week 29(N=54) | 4.06 [3.55 to 4.65]
  SC 20% individualized 1 Week- End of Study (N= 52) | 5.07 [4.48 to 5.73]

14. Secondary Outcome: Trough Levels of Anti-Hepatitis B Antibody
Time Frame: as for outcome 12
Population: Safety Analysis Set - sub-groups with data at relevant time points
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Study Epochs 1-4
Number analyzed (Participants) | 66
mIU/mL
  Pre-Study Medication- Epoch 1 Week 1 (N= 66) | 266.6 [232.3 to 305.9]
  IV 10% 3 Weeks- Epoch 1 Week 4 (N= 15) | 357.8 [312.2 to 410.1]
  IV 10% 3 Weeks- Epoch 1 Week 7 (N= 17) | 402.6 [333.4 to 486.0]
  IV 10% 3 Weeks- Epoch 1 Week 10 (N= 19) | 376.6 [315.7 to 449.3]
  IV 10% 3 Weeks- Epoch 1 Week 13 (N= 16) | 392.2 [310.4 to 495.6]
  IV 10% 4 Weeks- Epoch 1 Week 5 (N= 45) | 301.1 [266.2 to 340.5]
  IV 10% 4 Weeks- Epoch 1 Week 9 (N= 44) | 304.0 [271.0 to 341.0]
  IV 10% 4 Weeks- Epoch 1 Week 13 (N= 43) | 296.3 [266.0 to 330.2]
  SC 20% 145% IV 1 Week- Epoch 2 Week 5 (N= 29) | 463.7 [425.0 to 506.0]
  SC 20% 145% IV 1 Week- Epoch 2 Week 9 (N= 27) | 525.0 [478.1 to 576.5]
  SC 20% adjusted 1 Week- Epoch 3 Week 5 (N= 57) | 581.9 [533.4 to 634.9]
  SC 20% adjusted 1 Week- Epoch 3 Week 9 (N= 58) | 622.4 [579.8 to 668.1]
  SC 20% adjusted 1 Week- Epoch 4 Week 1 (N= 62) | 552.8 [509.7 to 599.6]
  SC 20% individualized 1 Week Epoch 4 Week 9(N= 58) | 434.4 [400.4 to 471.2]
  SC 20% individualized 1 Week Epoch 4 Week 17(N=53) | 444.5 [408.2 to 484.1]
  SC 20% individualized 1 Week Epoch 4 Week 29(N=54) | 389.2 [355.9 to 425.7]
  SC 20% individualized 1 Week- End of Study (N=56) | 403.1 [371.7 to 437.1]

15. Secondary Outcome: Pharmacokinetics Parameters for Immunoglobulin G (IgG): Area Under the Curve (AUC)
Description: The AUC between adjacent infusions will be calculated by the trapezoidal rule. Linear interpolation/extrapolation will be used to calculate the AUC for exact duration of the infusion intervals (21 or 28 days for IV administration and 7 days for SC administration). To allow for comparisons between Epochs 1, 2 and 4, AUC0-τ will be standardized for the infusion intervals (3 or 4 weeks vs. 1 week)
Time Frame: Epoch 1: 3 week IV interval: Weeks 10-13. Epoch 1: 4 week IV interval: Weeks 9-13. Epoch 2: Subcutaneous (SC) weeks 9-10. Epoch 4: SC weeks 17-18
Population: Safety Analysis Set - sub-groups with data at relevant time points
Measure: Geometric Mean (95% Confidence Interval); unit: g*days/L
Groups:
- Study Epoch 1: IGIV 10% Every 3 Weeks: Epoch 1 (13 weeks): Pharmacokinetic (PK) assessment at 2nd to last infusion (in all participants ≥12 years of age). Participants will be treated intravenously once every 3 weeks at same monthly equivalent dose as prior to the study. Immune globulin administered intravenously (IGIV)
- Study Epoch 1: IGIV 10% Every 4 Weeks: Epoch 1 (13 weeks): Pharmacokinetic (PK) assessment at 2nd to last infusion (in all participants ≥12 years of age). Participants will be treated intravenously once every 4 weeks at same monthly equivalent dose as prior to the study. Immune globulin administered intravenously (IGIV)
- Study Epoch 2: IGSC 20 %, 145 % of IGIV 10 %: Epoch 2 (12-16 weeks): PK assessment (in first 15 participants ≥12 years of age) at 9th infusion to determine adjusted dose for Epoch 3 and individually adapted dose for Epoch 4. Participants will be treated subcutaneously every 7 days at a dose of IGSC, 20% that is 145% of the weekly equivalent of the IV dose in Epoch 1. Immune globulin administered subcutaneously (IGSC)
- Study Epoch 4: IGSC 20 %, Individualized Dose: Epoch 4 (40 weeks): Participants will be treated subcutaneously once every week at the individually adapted dose determined in Epoch 3. PK assessment at 17th infusion. Immune globulin administered subcutaneously (IGSC)
Arm/Group | Study Epoch 1: IGIV 10% Every 3 Weeks | Study Epoch 1: IGIV 10% Every 4 Weeks | Study Epoch 2: IGSC 20 %, 145 % of IGIV 10 % | Study Epoch 4: IGSC 20 %, Individualized Dose
Number analyzed (Participants) | 16 | 38 | 18 | 60
g*days/L | 352.05 [319.74 to 387.63] | 410.40 [381.24 to 441.79] | 108.33 [97.60 to 120.24] | 115.21 [109.23 to 121.52]

16. Secondary Outcome: Pharmacokinetics Parameters for Immunoglobulin G (IgG): Dose Per Weight-adjusted Area Under the Curve (AUC)
Description: The AUC between adjacent infusions will be calculated by the trapezoidal rule. Linear interpolation/extrapolation will be used to calculate the AUC for exact duration of the infusion intervals (21 or 28 days for IV administration and 7 days for SC administration). To allow for comparisons between Epochs 1, 2 and 4, AUC0-τ will be standardized for the infusion intervals (3 or 4 weeks vs. 1 week) adjusted for the dose per weight.
Time Frame: as for outcome 15
Population: Safety Analysis Set - sub-groups with data at relevant time points
Measure: Geometric Mean (95% Confidence Interval); unit: (g*days/L)/(g/kg)
Groups:
- Study Epoch 4: IGSC 20 %, Individualized Dose: Epoch 4 (40 weeks): Participants will be treated subcutaneously once every week at the individually adapted dose determined in Epoch 3. PK assessment at 17th infusion. Immune globulin administered subcutaneously
Arm/Group | Study Epoch 1: IGIV 10% Every 3 Weeks | Study Epoch 1: IGIV 10% Every 4 Weeks | Study Epoch 2: IGSC 20 %, 145 % of IGIV 10 % | Study Epoch 4: IGSC 20 %, Individualized Dose
Number analyzed (Participants) | 16 | 38 | 18 | 60
(g*days/L)/(g/kg) | 606.99 [495.29 to 743.87] | 796.30 [715.36 to 886.40] | 472.50 [411.07 to 543.10] | 536.05 [495.58 to 579.82]

17. Secondary Outcome: Pharmacokinetics Parameters for Immunoglobulin G (IgG): Clearance (CL) for Immune Globulin Administered Intravenously (IGIV) and Apparent Clearance for Immune Globulin Administered Subcutaneously (IGSC)
Description: Clearance (CL) or apparent clearance (CL/F) for IV and SC administration, respectively, will be determined by the formula: CL or CL/F = (Dose (mg/kg)) / (AUC 0-τ). (F= bioavailability)
Time Frame: as for outcome 15
Population: Safety Analysis Set - sub-groups with data at relevant time point
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg/days
Arm/Group | Study Epoch 1: IGIV 10% Every 3 Weeks | Study Epoch 1: IGIV 10% Every 4 Weeks | Study Epoch 2: IGSC 20 %, 145 % of IGIV 10 % | Study Epoch 4: IGSC 20 %, Individualized Dose
Number analyzed (Participants) | 16 | 38 | 18 | 60
mL/kg/days | 1.65 [1.34 to 2.02] | 1.26 [1.13 to 1.40] | 2.12 [1.84 to 2.43] | 1.87 [1.72 to 2.02]

18. Secondary Outcome: Pharmacokinetics Parameters for Immunoglobulin G (IgG): Maximum Concentration (Cmax)
Description: The maximum concentration (Cmax) following administration of study drug (either immune globulin administered intravenously (IGIV) or immune globulin administered subcutaneously (IGSC).
Time Frame: as for outcome 15
Population: Safety Analysis Set - sub-groups with data at relevant time points
Measure: Geometric Mean (95% Confidence Interval); unit: g/L
Groups:
- Study Epoch 1: IGIV 10% Every 4 Week: Epoch 1 (13 weeks): Pharmacokinetic (PK) assessment at 2nd to last infusion (in all participants ≥12 years of age). Participants will be treated intravenously once every 4 weeks at same monthly equivalent dose as prior to the study. Immune globulin administered intravenously (IGIV)
Arm/Group | Study Epoch 1: IGIV 10% Every 3 Weeks | Study Epoch 1: IGIV 10% Every 4 Week | Study Epoch 2: IGSC 20 %, 145 % of IGIV 10 % | Study Epoch 4: IGSC 20 %, Individualized Dose
Number analyzed (Participants) | 16 | 38 | 18 | 60
g/L | 27.09 [24.30 to 30.19] | 24.85 [23.18 to 26.64] | 17.31 [15.11 to 19.82] | 19.31 [18.13 to 20.57]

19. Secondary Outcome: Pharmacokinetics Parameters for Immunoglobulin G (IgG): Time to Maximum Concentration (Tmax)
Description: The minimum time (Tmax) to reach the maximum concentration (Cmax)
Time Frame: as for outcome 15
Population: Safety Analysis Set - sub-groups with data at relevant time points
Measure: Geometric Mean (95% Confidence Interval); unit: hours (h)
Arm/Group | Study Epoch 1: IGIV 10% Every 3 Weeks | Study Epoch 1: IGIV 10% Every 4 Weeks | Study Epoch 2: IGSC 20 %, 145 % of IGIV 10 % | Study Epoch 4: IGSC 20 %, Individualized Dose
Number analyzed (Participants) | 16 | 38 | 18 | 60
hours (h) | 6.94 [3.96 to 12.17] | 5.84 [3.62 to 9.40] | 54.19 [36.28 to 80.92] | 78.68 [65.37 to 94.70]

20. Secondary Outcome: Pharmacokinetics Parameters for Immunoglobulin G (IgG): Minimum Concentration (Cmin)
Description: The minimum concentration (Cmax) following administration of study drug (either immune globulin administered intravenously (IGIV) or immune globulin administered subcutaneously (IGSC).
Time Frame: as for outcome 15
Population: Safety Analysis Set - sub-groups with data at relevant time points
Measure: Geometric Mean (95% Confidence Interval); unit: g/L
Arm/Group | Study Epoch 1: IGIV 10% Every 3 Weeks | Study Epoch 1: IGIV 10% Every 4 Weeks | Study Epoch 2: IGSC 20 %, 145 % of IGIV 10 % | Study Epoch 4: IGSC 20 %, Individualized Dose
Number analyzed (Participants) | 16 | 38 | 18 | 60
g/L | 12.03 [10.64 to 13.60] | 10.37 [9.50 to 11.33] | 13.85 [12.61 to 15.21] | 14.00 [13.14 to 14.91]

21. Secondary Outcome: Pharmacokinetics Parameters for Haemophilus Influenza B Antibody: Area Under the Curve (AUC)
Description: The AUC between adjacent infusions will be calculated by the trapezoidal rule . Linear interpolation/extrapolation will be used to calculate the AUC for exact duration of the infusion intervals (21 or 28 days for IV administration and 7 days for SC administration). To allow for comparisons between Epochs 1, 2 and 4, AUC 0-τ will be standardized for the infusion intervals (3 or 4 weeks vs. 1 week )
Time Frame: as for outcome 15
Population: Safety Analysis Set - sub-groups with data at relevant time points
Measure: Geometric Mean (95% Confidence Interval); unit: mg*days/L
Arm/Group | Study Epoch 1: IGIV 10% Every 3 Weeks | Study Epoch 1: IGIV 10% Every 4 Weeks | Study Epoch 2: IGSC 20 %, 145 % of IGIV 10 % | Study Epoch 4: IGSC 20 %, Individualized Dose
Number analyzed (Participants) | 16 | 37 | 18 | 59
mg*days/L | 80.79 [65.58 to 99.53] | 123.05 [93.36 to 162.18] | 29.51 [23.25 to 37.46] | 30.64 [26.29 to 35.72]

22. Secondary Outcome: Pharmacokinetics Parameters for Haemophilus Influenza B Antibody: Dose Per Weight-adjusted Area Under the Curve (AUC)
Description: The AUC between adjacent infusions will be calculated by the trapezoidal rule . Linear interpolation/extrapolation will be used to calculate the AUC for exact duration of the infusion intervals (21 or 28 days for IV administration and 7 days for SC administration). To allow for comparisons between Epochs 1, 2 and 4, AUC 0-τ will be standardized for the infusion intervals (3 or 4 weeks vs. 1 week) adjusted for the dose per weight.
Time Frame: as for outcome 15
Population: Safety Analysis Set - sub-groups with data at relevant time points
Measure: Geometric Mean (95% Confidence Interval); unit: (mg*days/L)/(g/kg)
Arm/Group | Study Epoch 1: IGIV 10% Every 3 Weeks | Study Epoch 1: IGIV 10% Every 4 Weeks | Study Epoch 2: IGSC 20 %, 145 % of IGIV 10 % | Study Epoch 4: IGSC 20 %, Individualized Dose
Number analyzed (Participants) | 16 | 37 | 18 | 59
(mg*days/L)/(g/kg) | 139.29 [110.89 to 174.97] | 239.99 [181.92 to 316.61] | 128.72 [96.65 to 171.42] | 141.78 [121.75 to 165.12]

23. Secondary Outcome: Pharmacokinetics Parameters for Haemophilus Influenza B Antibody: Clearance (CL) for Immune Globulin Administered Intravenously (IGIV) and Apparent Clearance (CL/F) for Immune Globulin Administered Subcutaneously
Description: Clearance (CL) or apparent clearance (CL/F) for IV and SC administration, respectively, will be determined by the formula: CL or CL/F = (Dose (mg/kg)) / (AUC 0- τ). (F= bioavailability)
Time Frame: as for outcome 15
Population: Safety Analysis Set - sub-groups with data at relevant time points
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg/days
Groups:
- Study Epoch 1: IGIV 10% Every 3 WeeksOverall Study Arm: Epoch 1 (13 weeks): Pharmacokinetic (PK) assessment at 2nd to last infusion (in all participants ≥12 years of age). Participants will be treated intravenously once every 3 weeks at same monthly equivalent dose as prior to the study. Immune globulin administered intravenously (IGIV)
- Study Epoch 2: IGSC 20%, 145% of IGIV 10%: Epoch 2 (12-16 weeks): PK assessment (in first 15 participants ≥12 years of age) at 9th infusion to determine adjusted dose for Epoch 3 and individually adapted dose for Epoch 4. Participants will be treated subcutaneously every 7 days at a dose of IGSC, 20% that is 145% of the weekly equivalent of the IV dose in Epoch 1. Immune globulin administered subcutaneously (IGSC)
- Study Epoch 4: IGSC 20%, Individualized Dose: Epoch 4 (40 weeks): Participants will be treated subcutaneously once every week at the individually adapted dose determined in Epoch 3. PK assessment at 17th infusion. Immune globulin administered subcutaneously
Arm/Group | Study Epoch 1: IGIV 10% Every 3 WeeksOverall Study Arm | Study Epoch 1: IGIV 10% Every 4 Weeks | Study Epoch 2: IGSC 20%, 145% of IGIV 10% | Study Epoch 4: IGSC 20%, Individualized Dose
Number analyzed (Participants) | 16 | 37 | 18 | 59
mL/kg/days | 7.18 [5.72 to 9.02] | 4.17 [3.16 to 5.50] | 7.77 [5.83 to 10.35] | 7.05 [6.06 to 8.21]

24. Secondary Outcome: Pharmacokinetics Parameters for Haemophilus Influenza B Antibody: Maximum Concentration (Cmax)
Description: as for outcome 18
Time Frame: as for outcome 15
Population: Safety Analysis Set - sub-groups with data at relevant time points
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Study Epoch 1: IGIV 10% Every 3 Weeks | Study Epoch 1: IGIV 10% Every 4 Weeks | Study Epoch 2: IGSC 20%, 145% of IGIV 10% | Study Epoch 4: IGSC 20 %, Individualized Dose
Number analyzed (Participants) | 16 | 37 | 18 | 59
mg/L | 6.31 [5.25 to 7.59] | 7.22 [5.75 to 9.05] | 4.40 [3.45 to 5.62] | 4.86 [4.16 to 5.68]

25. Secondary Outcome: Pharmacokinetics Parameters for Haemophilus Influenza B Antibody: Time to Maximum Concentration (Tmax)
Description: The minimum time (Tmax) to reach the maximum concentration (Cmax)
Time Frame: as for outcome 15
Population: Safety Analysis Set - sub-groups with data at relevant time points
Measure: Geometric Mean (95% Confidence Interval); unit: Hours (s)
Arm/Group | Study Epoch 1: IGIV 10% Every 3 Weeks | Study Epoch 1: IGIV 10% Every 4 Weeks | Study Epoch 2: IGSC 20 %, 145 % of IGIV 10 % | Study Epoch 4: IGSC 20 %, Individualized Dose
Number analyzed (Participants) | 16 | 37 | 18 | 59
Hours (s) | 3.11 [2.69 to 3.59] | 3.71 [2.69 to 5.12] | 70.67 [51.14 to 97.66] | 66.87 [56.22 to 79.53]

26. Secondary Outcome: Pharmacokinetics Parameters for Haemophilus Influenza B Antibody: Minimum Concentration (Cmin)
Description: as for outcome 20
Time Frame: as for outcome 15
Population: Safety Analysis Set - sub-groups with data at relevant time points
Measure: Median (95% Confidence Interval); unit: mg/L
Arm/Group | Study Epoch 1: IGIV 10% Every 3 Weeks | Study Epoch 1: IGIV 10% Every 4 Weeks | Study Epoch 2: IGSC 20%, 145% of IGIV 10% | Study Epoch 4: IGSC 20%, Individualized Dose
Number analyzed (Participants) | 16 | 37 | 18 | 59
mg/L | 2.82 [2.20 to 3.61] | 3.13 [2.31 to 4.26] | 3.97 [3.14 to 5.01] | 3.71 [3.15 to 4.37]

27. Secondary Outcome: Correction Factor to Determine the Individually Adapted Dose in Study 170904 Epoch 4 (Dose Adjustment Table)
Description: There is a high degree of variability in catabolism of immunoglobulin G (IgG) between individuals. To address this, trough levels immediately prior to the 9th weekly infusion in Epoch 3 were measured. The ratio of the measured trough levels on subcutaneous (SC) (Epoch 3) and intravenous (IV) administration (Epoch1) were compared to the expected trough level determined in Epoch 2. This was used to determine the Individually Adapted Dose to be used in Epoch 4. This was an interim study analysis.
Time Frame: 29 weeks
Population: Pharmacokinetics interim analysis set to determine the Individually Adapted Dose for Epoch 4
Measure: Number; unit: Correction factor
Arm/Group | Correction Factor
Number analyzed (Participants) | 15
Correction factor
  Trough Level Ratio: 0.93 or more | 1.16
  Trough Level Ratio: 0.94 | 1.14
  Trough Level Ratio: 0.95 to 0.96 | 1.12
  Trough Level Ratio: 0.97 to 0.98 | 1.11
  Trough Level Ratio: 0.99 to 1.01 | 1.10
  Trough Level Ratio: 1.02 to 1.04 | 1.09
  Trough Level Ratio: 1.05 to 1.08 | 1.08
  Trough Level Ratio: 1.09 to 1.13 | 1.07
  Trough Level Ratio: 1.14 to 1.19 | 1.06
  Trough Level Ratio: 1.20 to 1.26 | 1.05
  Trough Level Ratio: 1.27 to 1.33 | 1.04
  Trough Level Ratio: 1.34 to 1.40 | 1.03
  Trough Level Ratio: 1.41 to 1.47 | 1.02
  Trough Level Ratio: 1.48 to 1.55 | 1.01
  Trough Level Ratio: 1.56 to 1.63 | 1.00

28. Secondary Outcome: Number of Serious (SAEs) and Non-serious Adverse Events (AEs) (Including and Excluding Infections) Deemed Related to the Investigational Product Per Participant
Description: Number of related SAEs and AEs divided by number of participants
Time Frame: Up to 20 months per subject (throughout entire study)
Population: Safety Analysis Set
Measure: Number; unit: Adverse events per participant
Arm/Group | INTRAVENOUS 10% | SUBCUTANEOUS 20%
Number analyzed (Participants) | 77 | 74
Adverse events per participant
  Non-SAEs - Including infections | 1.039 | 2.122
  Non-SAEs - Excluding infections | 1.039 | 2.122
  SAEs - Including infections | 0.013 | 0
  SAEs - Excluding infections | 0.013 | 0

29. Secondary Outcome: Number of Serious (SAEs) and Non-serious Adverse Events (AEs) (Including and Excluding Infections) Deemed Related to the Investigational Product Per Infusion
Description: Number of related SAEs and AEs divided by number of subjects and divided by number of infusions
Time Frame: Up to 20 months per subject (throughout entire study)
Population: Safety Analysis Set
Measure: Number; unit: Adverse events per infusion
Units Other Than Participants: Infusions
Arm/Group | INTRAVENOUS 10% | SUBCUTANEOUS 20%
Number analyzed (Participants) | 77 | 74
Number analyzed (Infusions) | 324 | 4327
Adverse events per infusion
  Non-SAEs - Including Infections | 0.247 | 0.036
  Non-SAEs -Excluding Infections | 0.247 | 0.036
  SAEs - Including Infections | 0.003 | 0
  SAEs -Excluding Infections | 0.003 | 0

30. Secondary Outcome: Number of Serious (SAEs) and Non-serious Adverse Events (AEs) (Including and Excluding Infections) Regardless of Relationship to the Investigational Product Per Participant
Description: Number of all SAEs and AEs divided by number of participants
Time Frame: Up to 20 months per subject (throughout entire study)
Population: Safety Analysis Set
Measure: Number; unit: Adverse events per participant
Arm/Group | INTRAVENOUS 10% | SUBCUTANEOUS 20%
Number analyzed (Participants) | 77 | 74
Adverse events per participant
  Non-SAEs - Including infections | 3.325 | 9.014
  Non-SAEs - Excluding infections | 2.338 | 6.297
  SAEs - Including infections | 0.013 | 0.027
  SAEs - Excluding infections | 0.013 | 0.014

31. Secondary Outcome: Number of Serious (SAEs) and Non-serious Adverse Events (AEs) (Including and Excluding Infections) Regardless of Relationship to the Investigational Product Per Infusion
Description: Number of all SAEs and AEs divided by number of infusions
Time Frame: Up to 20 months per subject (throughout entire study)
Population: Safety Analysis Set
Measure: Number; unit: Adverse events per infusion
Units Other Than Participants: Infusions
Arm/Group | IGIV, 10% | Subcutaneous, 20%
Number analyzed (Participants) | 77 | 74
Number analyzed (Infusions) | 324 | 4327
Adverse events per infusion
  Non-SAEs - Including infections | 0.390 | 0.114
  Non-SAEs - Excluding infections | 0.296 | 0.079
  SAEs - including infections | 0.003 | 0.000
  SAEs - Excluding infections | 0.003 | 0.000

32. Secondary Outcome: Number of Adverse Events (AEs) (Including and Excluding Infections) That Begin During or Within 72 Hours of Completion of Infusion Per Participant
Description: Number of AEs that begin during or within 72 hours of completion of infusion divided by number of participants
Time Frame: Within 72 hours of completion of infusion
Population: Safety Analysis Set
Measure: Number; unit: Adverse events per participant
Arm/Group | Intravenous 10% | Subcutaneous 20%
Number analyzed (Participants) | 77 | 74
Adverse events per participant
  Non-SAEs - Including infections | 1.377 | 4.581
  Non-SAEs - Excluding infections | 1.260 | 3.703
  SAEs - Including infections | 0.013 | 0
  SAEs - Excluding infections | 0.013 | 0

33. Secondary Outcome: Number of Adverse Events (AEs) (Including and Excluding Infections) That Begin During or Within 72 Hours of Completion of Infusion Per Infusion
Description: Number of AEs that begin during or within 72 hours of completion of infusion divided by the number of infusions
Time Frame: Within 72 hours of completion of infusion
Population: Safety Analysis Set
Measure: Number; unit: Adverse events per infusion
Units Other Than Participants: Infusions
Arm/Group | Intravenous 10% | Subcutaneous 20%
Number analyzed (Participants) | 77 | 74
Number analyzed (Infusions) | 324 | 4327
Adverse events per infusion
  Non-SAEs - Including infections | 0.327 | 0.078
  Non-SAEs - Excluding infections | 0.299 | 0.063
  SAEs - Including infections | 0.003 | 0
  SAEs - Excluding infections | 0.003 | 0

34. Secondary Outcome: Number of Adverse Events (AEs) (Including and Excluding Infections) That Begin During or Within 24 Hours of Completion of Infusion Per Participant
Description: Number of AEs that begin during or within 24 hours of completion of infusion divided by number of participants
Time Frame: Within 24 hours of completion of infusion
Population: Safety Analysis Set
Measure: Number; unit: Adverse events per participant
Arm/Group | Intravenous 10% | Subcutaneous 20%
Number analyzed (Participants) | 77 | 74
Adverse events per participant
  Non-SAEs - Including infections | 0.961 | 3.365
  Non-SAEs - Excluding infections | 0.948 | 3.027
  SAEs - Including infections | 0 | 0
  SAEs - Excluding infections | 0 | 0

35. Secondary Outcome: Number of Adverse Events (AEs) (Including and Excluding Infections) That Begin During or Within 24 Hours of Completion of Infusion Per Infusion
Description: Number of AEs that begin during or within 24 hours of completion of infusion divided by number of infusions
Time Frame: Within 24 hours of completion of infusion
Population: Safety Analysis Set
Measure: Number; unit: Adverse events per infusion
Units Other Than Participants: Infusions
Arm/Group | Intravenous 10% | Subcutaneous 20%
Number analyzed (Participants) | 77 | 74
Number analyzed (Infusions) | 324 | 4327
Adverse events per infusion
  Non-SAEs - Including infections | 0.228 | 0.058
  Non-SAEs - Excluding infections | 0.225 | 0.052
  SAEs - Including infections | 0 | 0
  SAEs - Excluding infections | 0 | 0

36. Secondary Outcome: Number of Adverse Events (AEs) (Including and Excluding Infections) That Begin During or Within 1 Hour of Completion of Infusion Per Participant
Description: Number of AEs that begin during or within 1 hour of completion of infusion divided by number of participants
Time Frame: Within 1 hour of completion of infusion
Population: Safety Analysis Set
Measure: Number; unit: Adverse events per participant
Arm/Group | Intravenous 10% | Subcutaneous 20%
Number analyzed (Participants) | 77 | 74
Adverse events per participant
  Non-SAEs - Including infections | 0.662 | 1.865
  Non-SAEs - Excluding infections | 0.662 | 1.797
  SAEs - Including infections | 0 | 0
  SAEs - Excluding infections | 0 | 0

37. Secondary Outcome: Number of Adverse Events (AEs) (Including and Excluding Infections) That Begin During or Within 1 Hour of Completion of Infusion
Description: Number of AEs that begin during or within 1 hour of completion of infusion divided by number of infusions
Time Frame: Within 1 hour of completion of infusion
Population: Safety Analysis Set
Measure: Number; unit: Adverse events per infusion
Units Other Than Participants: Infusions
Arm/Group | Intravenous 10% | Subcutaneous 20%
Number analyzed (Participants) | 77 | 74
Number analyzed (Infusions) | 324 | 4327
Adverse events per infusion
  Non-SAEs - Including infections | 0.157 | 0.032
  Non-SAEs - Excluding infections | 0.157 | 0.031
  SAEs - Including infections | 0 | 0
  SAEs - Excluding infections | 0 | 0

38. Secondary Outcome: Causally Related and/or Temporally Associated Adverse Events (AEs) Per Infusion
Description: The total number of all AEs (including and excluding infections) that begin during infusion or within 72 hours of completion of an infusion ("temporally associated") plus the total number of AEs (including and excluding infections) starting more than 72 hours following the completion of an infusion determined by the investigator to be at least possibly related to the study drug("related"), divided by the total number of infusions
Time Frame: Within 72 hours post infusion for Temporally Associated AEs; End of each Study Epoch (Epoch 1, Epoch 2, Epoch 3, and Epoch 4) for Causally Related AEs
Population: Safety Analysis Set
Measure: Number; unit: Adverse events per infusion
Units Other Than Participants: Infusions
Arm/Group | Intravenous 10% | Subcutaneous 20%
Number analyzed (Participants) | 77 | 74
Number analyzed (Infusions) | 324 | 4327
Adverse events per infusion
  Non-SAEs - Including infections | 0.336 | 0.079
  Non-SAEs - Excluding infections | 0.309 | 0.064
  SAEs - Including infections | 0.003 | 0
  SAEs - Excluding infections | 0.003 | 0

39. Secondary Outcome: Percentage of Infusions Associated With One or More Local Non-serious Adverse Events (Non-SAEs)
Description: The number of infusions associated with local non-SAEs divided by the total number of infusions.
Time Frame: Up to 20 months (throughout entire study)
Population: Safety Analysis Set
Measure: Number; unit: Percent of infusions
Units Other Than Participants: Infusions
Arm/Group | Intravenous 10% | Subcutaneous 20%
Number analyzed (Participants) | 77 | 74
Number analyzed (Infusions) | 324 | 4327
Percent of infusions | 0.9 | 1.8

40. Secondary Outcome: Percentage of Participants Reporting One or More Local Non-serious Adverse Events (Non-SAEs)
Time Frame: Up to 20 months (throughout entire study)
Population: Safety Analysis Set
Measure: Number; unit: Percent of participants
Arm/Group | Intravenous 10% | Subcutaneous 20%
Number analyzed (Participants) | 77 | 74
Percent of participants | 3.9 | 31.1

41. Secondary Outcome: Number of Infusions for Which the Infusion Rate Was Reduced and/or the Infusion Was Interrupted or Stopped Due to Tolerability Concerns or AEs
Time Frame: Up to 20 months (throughout entire study)
Population: Safety Analysis Set
Measure: Number; unit: Infusions
Units Other Than Participants: Infusions
Arm/Group | Intravenous 10% | Subcutaneous 20%
Number analyzed (Participants) | 77 | 74
Number analyzed (Infusions) | 324 | 4327
Infusions
  Infusion rate reduced | 4 | 5
  Infusion interrupted | 5 | 2
  Infusion stopped | 0 | 1

42. Secondary Outcome: Percentage of Participants for Whom the Infusion Rate Was Reduced and/or the Infusion Was Interrupted or Stopped Due to Tolerability Concerns or AEs
Time Frame: Up to 20 months (throughout entire study)
Population: Safety Analysis Set
Measure: Number; unit: Percent of participants
Arm/Group | Intravenous 10% | Subcutaneous 20%
Number analyzed (Participants) | 77 | 74
Percent of participants
  Infusion rate reduced | 1.3 | 5.4
  Infusion interrupted | 6.5 | 1.4
  Infusion stopped | 0.0 | 1.4

43. Secondary Outcome: Percentage of Infusions Tolerated With Intravenous or Subcutaneous Administration
Description: An infusion will be deemed as tolerated unless one of the following occurs: 1. Any serious related AE(s) 2. Any non-serious local or systemic related AE(s) that prevent(s) completion of infusion 3. Any severe non-serious local or systemic related AE(s) that occur within 60 minutes of completion of the infusion
Time Frame: Up to 20 months (throughout entire study)
Population: Safety Analysis Set
Measure: Number; unit: Percent of infusions
Units Other Than Participants: Infusions
Arm/Group | Intravenous 10% | Subcutaneous 20%
Number analyzed (Participants) | 77 | 74
Number analyzed (Infusions) | 324 | 4327
Percent of infusions | 100 | 100

44. Secondary Outcome: Short Term Tolerance - Change in Systolic Blood Pressure: Immune Globulin Administered Intravenously (Human), 10% (IV 10%), Infusion 1
Description: Vital signs measured pre-infusion, during infusion, and post-infusion of Immune globulin administered intravenously (Human), 10% (IV 10%) was graded by the investigator and the sponsor using a 4-grade scale: mild (grade 1), moderate (grade 2), severe (grade 3) or life-threatening (grade 4) according to the U.S. Department of Health and Human Services, Food and Drug Administration, Center for Biologics Evaluation and Research; Guidance for Industry - Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, September2007. *Note 5th Grade (grade 0) added to scale to reflect within normal range.
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- Pre-Infusion Toxicity Grade 0: Normal Systolic Blood Pressure
- Pre-Infusion Toxicity Grade 1: Systolic Blood Pressure 141-150 mmHg
- Pre-Infusion Toxicity Grade 2: Systolic Blood Pressure 151-155 mmHg
- Pre-Infusion Toxicity Grade 3: Systolic Blood Pressure >155 mmHg
- Pre-Infusion Toxicity Grade 4: ER visit or hospitalization for malignant hypertension
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 72 | 2 | 3 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 61 | 1 | 1 | 0 | 0
  Maximum Post-Infusion Grade 1 | 10 | 1 | 1 | 0 | 0
  Maximum Post-Infusion Grade 2 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 1 | 0 | 1 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

45. Secondary Outcome: Short Term Tolerance - Change in Systolic Blood Pressure: Immune Globulin Administered Intravenously (Human), 10% (IV 10%), Infusion 2
Description: as for outcome 44
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 70 | 2 | 2 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 62 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 5 | 2 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 1 | 0 | 1 | 0 | 0
  Maximum Post-Infusion Grade 3 | 2 | 0 | 1 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

46. Secondary Outcome: Short Term Tolerance - Change in Systolic Blood Pressure: Immune Globulin Administered Intravenously (Human), 10% (IV 10%), Infusion 3
Description: as for outcome 44
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 69 | 2 | 3 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 59 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 9 | 2 | 2 | 0 | 0
  Maximum Post-Infusion Grade 2 | 1 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 1 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

47. Secondary Outcome: Short Term Tolerance - Change in Systolic Blood Pressure: Immune Globulin Administered Subcutaneously (Human), 20% (SC 20%), Infusion 1
Description: Vital signs measured pre-infusion, during infusion, and post-infusion of Immune globulin administered subcutaneously (Human), 20% (SC 20%) was graded by the investigator and the sponsor using a 4-grade scale: mild (grade 1), moderate (grade 2), severe (grade 3) or life-threatening (grade 4) according to the U.S. Department of Health and Human Services, Food and Drug Administration, Center for Biologics Evaluation and Research; Guidance for Industry - Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, September2007. *Note 5th Grade (grade 0) added to scale to reflect within normal range.
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 41 | 3 | 1 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 38 | 1 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 1 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 2 | 1 | 1 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 1 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

48. Secondary Outcome: Short Term Tolerance - Change in Systolic Blood Pressure: Immune Globulin Administered Subcutaneously (Human), 20% (SC 20%), Infusion 2
Description: as for outcome 47
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 37 | 3 | 0 | 1 | 0
Participants
  Maximum Post-Infusion Grade 0 | 35 | 2 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 2 | 1 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 0 | 1 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

49. Secondary Outcome: Short Term Tolerance - Change in Systolic Blood Pressure: Immune Globulin Administered Subcutaneously (Human), 20% (SC 20%), Infusion 3
Description: as for outcome 47
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 34 | 1 | 0 | 1 | 0
Participants
  Maximum Post-Infusion Grade 0 | 32 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 2 | 1 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 0 | 1 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

50. Secondary Outcome: Short Term Tolerance - Change in Diastolic Blood Pressure: Immune Globulin Administered Intravenously (Human), 10% (IV 10%), Infusion 1
Description: as for outcome 44
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- Pre-Infusion Toxicity Grade 0: Normal Diastolic Blood Pressure
- Pre-Infusion Toxicity Grade 1: Diastolic Blood Pressure 141-150 mmHg
- Pre-Infusion Toxicity Grade 2: Diastolic Blood Pressure 151-155 mmHg
- Pre-Infusion Toxicity Grade 3: Diastolic Blood Pressure >155 mmHg
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 72 | 1 | 3 | 1 | 0
Participants
  Maximum Post-Infusion Grade 0 | 69 | 0 | 1 | 0 | 0
  Maximum Post-Infusion Grade 1 | 2 | 0 | 2 | 0 | 0
  Maximum Post-Infusion Grade 2 | 0 | 1 | 0 | 1 | 0
  Maximum Post-Infusion Grade 3 | 1 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

51. Secondary Outcome: Short Term Tolerance - Change in Diastolic Blood Pressure: Immune Globulin Administered Intravenously (Human), 10% (IV 10%), Infusion 2
Description: as for outcome 44
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 71 | 2 | 1 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 67 | 0 | 1 | 0 | 0
  Maximum Post-Infusion Grade 1 | 3 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 1 | 2 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

52. Secondary Outcome: Short Term Tolerance - Change in Diastolic Blood Pressure: Immune Globulin Administered Intravenously (Human), 10% (IV 10%), Infusion 3
Description: as for outcome 44
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 71 | 3 | 0 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 69 | 1 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 1 | 2 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 1 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

53. Secondary Outcome: Short Term Tolerance - Change in Diastolic Blood Pressure: Immune Globulin Administered Subcutaneously (Human), 20% (SC 20%), Infusion 1
Description: as for outcome 47
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 42 | 3 | 0 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 41 | 1 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 0 | 1 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 1 | 1 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

54. Secondary Outcome: Short Term Tolerance - Change in Diastolic Blood Pressure: Immune Globulin Administered Subcutaneously (Human), 20% (SC 20%), Infusion 2
Description: as for outcome 47
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 39 | 1 | 1 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 37 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 2 | 1 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 1 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

55. Secondary Outcome: Short Term Tolerance - Change in Diastolic Blood Pressure: Immune Globulin Administered Subcutaneously (Human), 20% (SC 20%), Infusion 3
Description: as for outcome 47
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 35 | 0 | 1 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 35 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 0 | 0 | 1 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

56. Secondary Outcome: Short Term Tolerance - Change in Heart Rate (Pulse): Immune Globulin Administered Intravenously (Human), 10% (IV 10%), Infusion 1
Description: as for outcome 44
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- Pre-Infusion Toxicity Grade 0: Normal Heart Rate (Pulse)
- Pre-Infusion Toxicity Grade 1: Heart Rate (Pulse): Either Bradycardia (50 - 54 beats per minute) OR Tachycardia (101 - 115 beats per minute)
- Pre-Infusion Toxicity Grade 2: Heart Rate (Pulse): Either Bradycardia (45 - 49 beats per minute) OR Tachycardia (116 - 130 beats per minute)
- Pre-Infusion Toxicity Grade 3: Heart Rate (Pulse): Either Bradycardia (< 45 beats per minute) OR Tachycardia (> 130 beats per minute)
- Pre-Infusion Toxicity Grade 4: Heart Rate (Pulse): Either Bradycardia (ER visit or hospitalization for arrhythmia) OR Tachycardia (ER visit or hospitalization for arrhythmia)
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 71 | 4 | 1 | 1 | 0
Participants
  Maximum Post-Infusion Grade 0 | 61 | 3 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 8 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 2 | 1 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 1 | 1 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

57. Secondary Outcome: Short Term Tolerance - Change in Heart Rate (Pulse): Immune Globulin Administered Intravenously (Human), 10% (IV 10%), Infusion 2
Description: as for outcome 44
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 66 | 6 | 2 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 53 | 3 | 1 | 0 | 0
  Maximum Post-Infusion Grade 1 | 9 | 2 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 4 | 0 | 1 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 1 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

58. Secondary Outcome: Short Term Tolerance - Change in Heart Rate (Pulse): Immune Globulin Administered Intravenously (Human), 10% (IV 10%), Infusion 3
Description: as for outcome 44
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 66 | 5 | 3 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 55 | 1 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 9 | 2 | 1 | 0 | 0
  Maximum Post-Infusion Grade 2 | 2 | 2 | 2 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

59. Secondary Outcome: Short Term Tolerance - Change in Heart Rate (Pulse): Immune Globulin Administered Subcutaneously (Human), 20% (SC 20%), Infusion 1
Description: as for outcome 47
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 43 | 2 | 0 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 40 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 1 | 2 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 2 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

60. Secondary Outcome: Short Term Tolerance - Change in Heart Rate (Pulse): Immune Globulin Administered Subcutaneously (Human), 20% (SC 20%), Infusion 2
Description: as for outcome 47
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 39 | 2 | 0 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 36 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 2 | 2 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 1 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

61. Secondary Outcome: Short Term Tolerance - Change in Heart Rate (Pulse): Immune Globulin Administered Subcutaneously (Human), 20% (SC 20%), Infusion 3
Description: as for outcome 47
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 33 | 3 | 0 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 32 | 2 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 1 | 1 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

62. Secondary Outcome: Short Term Tolerance - Change in Respiratory Rate: Immune Globulin Administered Intravenously (Human), 10% (IV 10%), Infusion 1
Description: as for outcome 44
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- Pre-Infusion Toxicity Grade 0: Normal Respiratory Rate
- Pre-Infusion Toxicity Grade 1: Respiratory Rate: 17 - 20 breaths per minute
- Pre-Infusion Toxicity Grade 2: Respiratory Rate: 21 - 25 breaths per minute
- Pre-Infusion Toxicity Grade 3: Respiratory Rate: > 25 breaths per minute
- Pre-Infusion Toxicity Grade 4: Intubation
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 39 | 35 | 3 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 32 | 5 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 7 | 28 | 1 | 0 | 0
  Maximum Post-Infusion Grade 2 | 0 | 2 | 2 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

63. Secondary Outcome: Short Term Tolerance - Change in Respiratory Rate: Immune Globulin Administered Intravenously (Human), 10% (IV 10%), Infusion 2
Description: as for outcome 44
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 46 | 23 | 3 | 2 | 0
Participants
  Maximum Post-Infusion Grade 0 | 35 | 2 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 11 | 19 | 1 | 0 | 0
  Maximum Post-Infusion Grade 2 | 0 | 1 | 2 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 1 | 0 | 2 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

64. Secondary Outcome: Short Term Tolerance - Change in Respiratory Rate: Immune Globulin Administered Intravenously (Human), 10% (IV 10%), Infusion 3
Description: as for outcome 44
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 38 | 32 | 2 | 2 | 0
Participants
  Maximum Post-Infusion Grade 0 | 32 | 4 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 6 | 26 | 2 | 0 | 0
  Maximum Post-Infusion Grade 2 | 0 | 2 | 0 | 1 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 0 | 1 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

65. Secondary Outcome: Short Term Tolerance - Change in Respiratory Rate: Immune Globulin Administered Subcutaneously (Human), 20% (SC 20%), Infusion 1
Description: as for outcome 47
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 27 | 18 | 0 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 18 | 1 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 9 | 17 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

66. Secondary Outcome: Short Term Tolerance - Change in Respiratory Rate: Immune Globulin Administered Subcutaneously (Human), 20% (SC 20%), Infusion 2
Description: as for outcome 47
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 22 | 19 | 0 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 18 | 1 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 4 | 18 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

67. Secondary Outcome: Short Term Tolerance - Change in Respiratory Rate: Immune Globulin Administered Subcutaneously (Human), 20% (SC 20%), Infusion 3
Description: as for outcome 47
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 18 | 17 | 1 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 13 | 6 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 5 | 11 | 1 | 0 | 0
  Maximum Post-Infusion Grade 2 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

68. Secondary Outcome: Short Term Tolerance - Change in Body Temperature: Immune Globulin Administered Intravenously (Human), 10% (IV 10%), Infusion 1
Description: as for outcome 47
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- Pre-Infusion Toxicity Grade 0: Normal Body temperature
- Pre-Infusion Toxicity Grade 1: Body Temperature, Fever (°C) of: 38.0 - 38.4
- Pre-Infusion Toxicity Grade 2: Body Temperature, Fever (°C) of: 38.5 - 38.9
- Pre-Infusion Toxicity Grade 3: Body Temperature, Fever (°C) of: 39.0 - 40
- Pre-Infusion Toxicity Grade 4: Body Temperature, Fever (°C) of: > 40
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 77 | 0 | 0 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 77 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

69. Secondary Outcome: Short Term Tolerance - Change in Body Temperature: Immune Globulin Administered Intravenously (Human), 10% (IV 10%), Infusion 2
Description: as for outcome 44
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 74 | 0 | 0 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 73 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 1 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

70. Secondary Outcome: Short Term Tolerance - Change in Body Temperature: Immune Globulin Administered Intravenously (Human), 10% (IV 10%), Infusion 3
Description: as for outcome 44
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 74 | 0 | 0 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 72 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 2 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

71. Secondary Outcome: Short Term Tolerance - Change in Body Temperature: Immune Globulin Administered Subcutaneously (Human), 20% (SC 20%), Infusion 1
Description: as for outcome 47
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 45 | 0 | 0 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 45 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

72. Secondary Outcome: Short Term Tolerance - Change in Body Temperature: Immune Globulin Administered Subcutaneously (Human), 20% (SC 20%), Infusion 2
Description: as for outcome 47
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 41 | 0 | 0 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 41 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

73. Secondary Outcome: Short Term Tolerance - Change in Body Temperature: Immune Globulin Administered Subcutaneously (Human), 20% (SC 20%), Infusion 3
Description: as for outcome 47
Time Frame: Within 30 minutes pre-infusion, during infusion and within 30 minutes post infusion
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Infusion Toxicity Grade 0 | Pre-Infusion Toxicity Grade 1 | Pre-Infusion Toxicity Grade 2 | Pre-Infusion Toxicity Grade 3 | Pre-Infusion Toxicity Grade 4
Number analyzed (Participants) | 36 | 0 | 0 | 0 | 0
Participants
  Maximum Post-Infusion Grade 0 | 36 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 1 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 2 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 3 | 0 | 0 | 0 | 0 | 0
  Maximum Post-Infusion Grade 4 | 0 | 0 | 0 | 0 | 0

74. Secondary Outcome: Number of Participants With Laboratory Confirmed Hemolysis That Occurred Following Investigational Product Administration
Description: Laboratory tests for confirmation of potential hemolysis include Coomb's test, haptoglobin, free hemoglobin, reticulocyte count, lactate dehydrogenase (LDH), and urine hemosiderin.
Time Frame: Epoch 1: 3 week IV interval- weeks 0, 10. Epoch 1: 4 week IV interval- weeks 0, 9. Epoch 3: Subcutaneous (SC) week 9. Epoch 4: SC weeks 17, 18, 40
Population: Safety Analysis Set
Measure: Number; unit: Participants
Arm/Group | Intravenous 10% | Subcutaneous 20%
Number analyzed (Participants) | 77 | 74
Participants | 0 | 0

75. Secondary Outcome: Quality of Life- Pediatric Quality of Life Inventory^TM (PEDS-QL^TM) (Observer: Parent) for the Age Group 2 to 7 Years
Description: The Peds-QL is a generic Health-Related Quality of Life (HR QoL) instrument designed specifically for a pediatric population. It captures the following domains: general health/activities, feelings/emotional, social functioning, school functioning. Higher scores indicate better quality of life (QoL) for all domains of the Peds-QL. This modular instrument uses a 5-point scale: from 0 (never) to 4 (almost always). Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. 4 dimensions (physical, emotional, social, & school functioning) are scored. 2 summary scores (Psychosocial Health Summary, and Physical Health Summary) are presented, along with a total score.
Time Frame: Up to 20 months (throughout entire study)
Population: Safety Analysis Set (subset of participants aged 2 to 7 years)
Measure: Median (95% Confidence Interval); unit: Score on a scale
Groups:
- Start of Study Epoch 1; End of Study Epoch 1: Epoch 1 (13 weeks): Participants will be treated intravenously once every 3 or 4 weeks at same monthly equivalent dose as prior to the study.
- End of Study Epoch 3: Epoch 3 (12 weeks): Participants will be treated subcutaneously every 7 days using the adjusted dose determined in Epoch 2. The individually adapted dose for use in Epoch 4 will also be determined.
- End of Study Epoch 4: Epoch 4 (40 weeks): Participants will be treated subcutaneously once every week at the individually adapted dose determined in Epoch 3.
- Change End Epoch 1 to End Epoch 3: Epoch 1 (13 weeks): Participants will be treated intravenously once every 3 or 4 weeks at same monthly equivalent dose as prior to the study. Epoch 3 (12 weeks): Participants will be treated subcutaneously every 7 days using the adjusted dose determined in Epoch 2. The individually adapted dose for use in Epoch 4 will also be determined.
- Change End Epoch 1 to End Epoch 4: Epoch 1 (13 weeks): Participants will be treated intravenously once every 3 or 4 weeks at same monthly equivalent dose as prior to the study. Epoch 4 (40 weeks): Participants will be treated subcutaneously once every week at the individually adapted dose determined in Epoch 3.
Arm/Group | Start of Study Epoch 1 | End of Study Epoch 1 | End of Study Epoch 3 | End of Study Epoch 4 | Change End Epoch 1 to End Epoch 3 | Change End Epoch 1 to End Epoch 4
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
Score on a scale
  Physical Functioning | 95.31 [68.75 to 100.00] | 93.75 [56.25 to 100.00] | 96.88 [62.50 to 100.00] | 92.19 [75.00 to 100.00] | 1.56 [-3.13 to 9.38] | 1.56 [-12.50 to 18.75]
  Emotional Functioning | 95.00 [70.00 to 95.00] | 85.00 [50.00 to 95.00] | 82.50 [60.00 to 100.00] | 77.50 [55.00 to 85.00] | 0.00 [-5.00 to 10.00] | -2.50 [-20.00 to 10.00]
  Social Functioning | 95.00 [65.00 to 100.00] | 95.00 [25.00 to 100.00] | 97.50 [25.00 to 100.00] | 87.50 [50.00 to 100.00] | 0.00 [-5.00 to 10.00] | 0.00 [-15.00 to 25.00]
  School Functioning | 85.00 [55.00 to 100.00] | 75.00 [30.00 to 83.33] | 81.67 [40.00 to 100.00] | 67.50 [25.00 to 91.67] | 7.50 [0.00 to 25.00] | -5.00 [-10.00 to 8.33]
  Psychosocial Health Summary | 91.67 [65.00 to 98.08] | 83.33 [38.33 to 92.31] | 84.17 [41.67 to 100.00] | 77.50 [46.67 to 90.38] | 2.50 [0.00 to 11.67] | -3.33 [-8.33 to 8.33]
  Physical Health Summary | 95.31 [68.75 to 100.00] | 93.75 [56.25 to 100.00] | 96.88 [62.50 to 100.00] | 92.19 [75.00 to 100.00] | 1.56 [-3.13 to 9.38] | 1.56 [-12.50 to 18.75]
  Total Score | 92.93 [69.57 to 98.81] | 86.96 [59.78 to 94.05] | 88.04 [60.87 to 100.00] | 82.61 [60.87 to 94.05] | 1.63 [0.00 to 10.87] | 0.00 [-5.43 to 4.35]

76. Secondary Outcome: Quality of Life- PEDS-QL^TM (Observer: Participant) for the Age Group 8 to 13 Years of Age
Description: as for outcome 75
Time Frame: Up to 20 months (throughout entire study)
Population: Safety Analysis Set participants aged 8 to 13 with scores at each respective time point.
Measure: Median (95% Confidence Interval); unit: Score on a scale
Groups:
- Start of Epoch 1; End of Epoch 1: Epoch 1 (13 weeks): Participants will be treated intravenously once every 3 or 4 weeks at same monthly equivalent dose as prior to the study.
- End of Epoch 3: Epoch 3 (12 weeks): Participants will be treated subcutaneously every 7 days using the adjusted dose determined in Epoch 2. The individually adapted dose for use in Epoch 4 will also be determined.
- End of Epoch 4: Epoch 4 (40 weeks): Participants will be treated subcutaneously once every week at the individually adapted dose determined in Epoch 3.
- Change End of Epoch 1 to End of Epoch 3: Epoch 1 (13 weeks): Participants will be treated intravenously once every 3 or 4 weeks at same monthly equivalent dose as prior to the study. Epoch 3 (12 weeks): Participants will be treated subcutaneously every 7 days using the adjusted dose determined in Epoch 2. The individually adapted dose for use in Epoch 4 will also be determined.
- Change End of Epoch 1 to End of Epoch 4: Epoch 1 (13 weeks): Participants will be treated intravenously once every 3 or 4 weeks at same monthly equivalent dose as prior to the study. Epoch 4 (40 weeks): Participants will be treated subcutaneously once every week at the individually adapted dose determined in Epoch 3.
Arm/Group | Start of Epoch 1 | End of Epoch 1 | End of Epoch 3 | End of Epoch 4 | Change End of Epoch 1 to End of Epoch 3 | Change End of Epoch 1 to End of Epoch 4
Number analyzed (Participants) | 14 | 15 | 15 | 14 | 15 | 14
Score on a scale
  Physical Functioning | 89.06 [81.25 to 100.00] | 90.63 [78.13 to 100.00] | 87.50 [75.00 to 100.00] | 93.75 [71.88 to 100.00] | 0.00 [-3.13 to 9.38] | 6.25 [0.00 to 15.63]
  Emotional Functioning | 87.50 [75.00 to 100.00] | 80.00 [70.00 to 90.00] | 80.00 [70.00 to 95.00] | 87.50 [65.00 to 95.00] | 0.00 [-5.00 to 5.00] | 10.00 [-5.00 to 15.00]
  Social Functioning | 87.50 [80.00 to 100.00] | 95.00 [80.00 to 100.00] | 95.00 [85.00 to 100.00] | 95.00 [85.00 to 100.00] | 0.00 [0.00 to 5.00] | 0.00 [0.00 to 5.00]
  School Functioning | 75.00 [55.00 to 90.00] | 80.00 [60.00 to 85.00] | 75.00 [55.00 to 85.00] | 70.00 [55.00 to 85.00] | 0.00 [-10.00 to 10.00] | -2.50 [-15.00 to 10.00]
  Psychosocial Health Summary | 80.83 [76.67 to 91.67] | 83.33 [71.67 to 91.67] | 81.67 [75.00 to 93.33] | 81.67 [78.33 to 91.67] | 0.00 [-3.33 to 8.33] | 3.33 [-1.67 to 10.00]
  Physical Health Summary | 89.06 [81.25 to 100.00] | 90.63 [78.13 to 100.00] | 87.50 [75.00 to 100.00] | 93.75 [71.88 to 100.00] | 0.00 [-3.13 to 9.38] | 6.25 [0.00 to 15.63]
  Total Score | 86.41 [82.61 to 94.57] | 89.13 [69.57 to 91.30] | 81.52 [76.09 to 93.48] | 85.87 [79.35 to 92.39] | 1.09 [-1.09 to 7.61] | 2.17 [-3.26 to 10.87]

77. Secondary Outcome: Quality of Life- Short-Form 36v2 (SF-36v2) for the Age Group 14 Years and Older
Description: The PCS is a summary scale of the dimensions physical functioning, role physical, bodily pain, and general health. The component score is normalized to a standard population. Scores range from 0 to 100 with higher scores representing better health. There is no total overall score; scoring is done for both sub-scores and summary scores.
Time Frame: Up to 20 months (throughout entire study)
Population: Safety Analysis Set participants aged 14 years and older with scores at each respective time point.
Measure: Median (95% Confidence Interval); unit: Scores on a scale
Arm/Group | START OF STUDY EPOCH 1 | END OF STUDY EPOCH 1 | END OF STUDY EPOCH 3 | END OF STUDY EPOCH 4 | CHANGE END EPOCH 1 TO END EPOCH 3 | CHANGE END EPOCH 1 TO END EPOCH 4
Number analyzed (Participants) | 56 | 53 | 49 | 48 | 49 | 48
Scores on a scale
  Physical Functioning | 48.61 [46.51 to 52.82] | 52.82 [44.41 to 54.93] | 50.72 [48.61 to 52.82] | 50.72 [46.51 to 54.93] | 0.00 [-2.10 to 0.00] | 0.00 [-2.10 to 2.10]
  Role-Physical | 44.61 [37.26 to 49.51] | 42.16 [37.26 to 51.96] | 49.51 [42.16 to 54.40] | 47.06 [44.61 to 51.96] | 2.45 [0.00 to 4.90] | 2.45 [0.00 to 4.90]
  Bodily Pain | 43.95 [41.41 to 51.13] | 45.64 [37.18 to 50.29] | 50.29 [41.83 to 51.13] | 46.06 [41.83 to 51.13] | 4.23 [0.00 to 4.65] | 0.00 [0.00 to 4.65]
  General Health | 38.63 [33.87 to 41.02] | 41.02 [33.87 to 44.83] | 38.63 [36.25 to 45.78] | 38.63 [36.25 to 45.78] | 0.95 [-1.43 to 2.38] | 0.72 [-2.38 to 2.38]
  Vitality | 42.72 [39.60 to 48.97] | 42.72 [36.48 to 48.97] | 45.85 [39.60 to 52.09] | 48.97 [42.72 to 52.09] | 3.12 [0.00 to 3.12] | 1.56 [0.00 to 6.24]
  Social Functioning | 45.94 [40.49 to 51.40] | 45.94 [40.49 to 51.40] | 51.40 [45.94 to 51.40] | 51.40 [45.94 to 56.85] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 5.45]
  Role-Emotional | 51.99 [44.22 to 55.88] | 55.88 [48.10 to 55.88] | 51.99 [48.10 to 55.88] | 53.94 [44.22 to 55.88] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Mental Health | 50.01 [47.19 to 52.82] | 52.82 [47.19 to 55.64] | 50.01 [47.19 to 52.82] | 52.82 [50.01 to 55.64] | 0.00 [-2.82 to 2.82] | 1.41 [-2.82 to 2.82]
  Physical Component Summary | 41.57 [38.01 to 47.02] | 39.93 [37.57 to 47.98] | 46.13 [43.00 to 50.84] | 46.07 [42.38 to 49.25] | 1.22 [-0.51 to 3.29] | 0.89 [-0.37 to 2.49]
  Mental Component Summary | 49.92 [45.53 to 51.78] | 49.45 [46.87 to 53.58] | 49.70 [46.37 to 54.06] | 51.59 [48.03 to 54.35] | 0.57 [-2.17 to 2.39] | 1.31 [-3.69 to 4.40]

78. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM) - 2 to 12 Years Old
Description: TSQM; for the age group 2 to 12 years the observer will be a parent. Treatment Satisfaction Questionnaire for Medication (TSQM) is a global satisfaction scale used to assess the overall level of participant's satisfaction or dissatisfaction with their medications. The following 3 domain were included: effectiveness, convenience, and global satisfaction. The score of each of the 3 domains is based on an algorithm to create a score of 0 to 100. Higher score indicated greater satisfaction in that domain.
Time Frame: Up to 20 months per subject (throughout entire study)
Population: Safety Analysis Set - participants aged 2-12 years old with data (scores) at relevant time points
Measure: Median (95% Confidence Interval); unit: Score on a scale
Arm/Group | Start of Epoch 1 | End of Epoch 1 | End of Epoch 3 | End of Epoch 4 | Change End of Epoch 1 to End of Epoch 3 | Change End of Epoch 1 to End of Epoch 4
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16
Score on a scale
  Effectiveness | 83.33 [77.78 to 100.00] | 88.89 [83.33 to 100.00] | 83.33 [66.67 to 100.00] | 91.67 [72.22 to 100.00] | 0.00 [-11.11 to 0.00] | 0.00 [-5.56 to 5.56]
  Convenience | 75.00 [55.56 to 88.89] | 72.22 [66.67 to 83.33] | 80.56 [77.78 to 100.00] | 77.78 [77.78 to 94.44] | 5.56 [0.00 to 27.78] | 5.56 [0.00 to 16.67]
  Global Satisfaction | 85.71 [78.57 to 100.00] | 92.86 [71.43 to 100.00] | 100.00 [71.43 to 100.00] | 89.29 [71.43 to 100.00] | 0.00 [0.00 to 7.14] | 0.00 [0.00 to 7.14]

79. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM) - 13 Years and Older
Description: TSQM; for the age group 13 years and older the observer will be the participant. Treatment Satisfaction Questionnaire for Medication (TSQM) is a global satisfaction scale used to assess the overall level of participant's satisfaction or dissatisfaction with their medications. The following 3 domain were included: effectiveness, convenience, and global satisfaction. The score of each of the 3 domains is based on an algorithm to create a score of 0 to 100. Higher score indicated greater satisfaction in that domain.
Time Frame: Up to 20 months per subject (throughout entire study)
Population: Safety Analysis Set - participants aged 13 years and older with data (scores) at relevant time points
Measure: Median (95% Confidence Interval); unit: Score on a scale
Arm/Group | Start of Epoch 1 | End of Epoch 1 | End of Epoch 3 | End of Epoch 4 | Change End of Epoch 1 to End of Epoch 3 | Change End of Epoch 1 to End of Epoch 4
Number analyzed (Participants) | 61 | 58 | 54 | 53 | 54 | 53
Score on a scale
  Effectiveness | 77.78 [72.22 to 83.33] | 80.56 [72.22 to 88.89] | 83.33 [77.78 to 88.89] | 83.33 [77.78 to 88.89] | 0.00 [0.00 to 5.56] | 0.00 [0.00 to 5.56]
  Convenience | 66.67 [61.11 to 77.78] | 66.67 [55.56 to 72.22] | 83.33 [72.22 to 83.33] | 83.33 [77.78 to 88.89] | 11.11 [5.56 to 16.67] | 11.11 [5.56 to 16.67]
  Global Satisfaction | 85.71 [78.57 to 92.86] | 85.71 [78.57 to 92.86] | 92.86 [78.57 to 92.86] | 92.86 [85.71 to 92.86] | 0.00 [0.00 to 7.14] | 0.00 [0.00 to 7.14]

80. Secondary Outcome: Life Quality Index - 2 to 12 Years Old
Description: For the age group 2 to 12 years the respondent will be a parent. Each of the four domains has a separate score, each has a different range as follows: Treatment Interference Score Range: 6-42, Therapy-related Problems Score Range: 4-28, Therapy Setting Score Range: 3-21, Cost Score Range: 2-14. Higher scores represent more satisfaction with various aspects of treatment.
Time Frame: Up to 20 months (throughout entire study)
Population: Safety Analysis Set - participants aged 2-12 years old with data (scores) at relevant time points
Measure: Median (95% Confidence Interval); unit: Score on a scale
Arm/Group | Start of Epoch 1 | End of Epoch 1 | End of Epoch 3 | End of Epoch 4 | Change End of Epoch 1 to End of Epoch 3 | Change End of Epoch 1 to End of Epoch 4
Number analyzed (Participants) | 16 | 16 | 15 | 16 | 15 | 16
Score on a scale
  Treatment Interference | 32.0 [27.0 to 40.0] | 31.0 [30.0 to 41.0] | 35.0 [31.0 to 39.0] | 34.5 [30.0 to 39.0] | 0.0 [-2.0 to 5.0] | -0.5 [-2.0 to 9.0]
  Therapy-related Problems | 23.0 [20.0 to 24.0] | 23.0 [22.0 to 26.0] | 22.0 [20.0 to 24.0] | 21.5 [21.0 to 25.0] | 0.0 [-2.0 to 0.0] | -1.0 [-3.0 to 0.0]
  Therapy Settings | 18.0 [17.0 to 21.0] | 18.0 [16.0 to 20.0] | 19.0 [18.0 to 21.0] | 20.0 [17.0 to 21.0] | 0.0 [0.0 to 3.0] | 1.0 [-1.0 to 3.0]
  Costs | 9.0 [8.0 to 11.0] | 11.0 [10.0 to 13.0] | 11.0 [11.0 to 12.0] | 10.5 [9.0 to 13.0] | 1.0 [0.0 to 2.0] | -0.5 [-1.0 to 2.0]

81. Secondary Outcome: Life Quality Index - 13 Years and Older
Description: For the age group 13 years and older the respondent will be the participant. Each of the four domains has a separate score, each has a different range as follows: Treatment Interference Score Range: 6-42, Therapy-related Problems Score Range: 4-28, Therapy Setting Score Range: 3-21, Cost Score Range: 2-14. Higher scores represent more satisfaction with various aspects of treatment.
Time Frame: Up to 20 months per subject (throughout entire study)
Population: Safety Analysis Set - participants aged 13 years and older with data (scores) at relevant time points
Measure: Median (95% Confidence Interval); unit: Score on a scale
Arm/Group | Start of Epoch 1 | End of Epoch 1 | End of Epoch 3 | End of Epoch 4 | Change End of Epoch 1 to End of Epoch 3 | Change End of Epoch 1 to End of Epoch 4
Number analyzed (Participants) | 61 | 58 | 54 | 52 | 54 | 52
Score on a scale
  Treatment Interference | 34.0 [30.0 to 37.0] | 34.5 [32.0 to 36.0] | 37.0 [35.0 to 39.0] | 38.5 [34.0 to 40.0] | 1.0 [0.0 to 4.0] | 3.0 [0.0 to 5.0]
  Therapy-related Problems | 23.0 [22.0 to 24.0] | 22.5 [21.0 to 24.0] | 24.0 [22.0 to 25.0] | 24.0 [23.0 to 25.0] | 0.0 [-1.0 to 2.0] | 1.0 [-1.0 to 2.0]
  Therapy Settings | 18.0 [16.0 to 19.0] | 17.0 [16.0 to 18.0] | 20.0 [19.0 to 20.0] | 20.0 [19.0 to 21.0] | 1.0 [0.0 to 3.0] | 2.0 [0.0 to 3.0]
  Costs | 8.0 [7.0 to 10.0] | 10.0 [9.0 to 10.0] | 11.5 [10.0 to 13.0] | 13.0 [11.0 to 14.0] | 1.0 [0.0 to 2.0] | 1.5 [1.0 to 3.0]

ADVERSE EVENTS:
Time Frame: Throughout the 4 Study Epochs. Epoch 1: 13 weeks. Epoch 2: 12-16 weeks Epoch 3: 12 weeks Epoch 4: 40 weeks
Arm/Group | Study Epoch 1: Intravenous 10% Treatment | Study Epochs 2-4: Subcutaneous 20% Treatment
Serious Adverse Events (participants affected / at risk) | 1/77 | 2/74
Other Adverse Events (participants affected / at risk) | 46/77 | 59/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Epoch 1: Intravenous 10% Treatment (N=77) | Study Epochs 2-4: Subcutaneous 20% Treatment (N=74)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Lung adenocarcinima (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Epoch 1: Intravenous 10% Treatment (N=77) | Study Epochs 2-4: Subcutaneous 20% Treatment (N=74)
Sinusitis (Infections and infestations) | 7 (8) | 18 (29)
Acute sinusitis (Infections and infestations) | 6 (8) | 15 (22)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 14 (21)
Infusion site pain (General disorders) | 0 (0) | 14 (34)
Headache (Nervous system disorders) | 23 (44) | 12 (54)
Nausea (Gastrointestinal disorders) | 6 (11) | 11 (21)
Bronchitis (Nervous system disorders) | 3 (3) | 11 (14)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 8 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (9)
Infusion site erythema (General disorders) | 0 (0) | 8 (23)
Fatigue (General disorders) | 5 (6) | 7 (12)
Nasopharyngitis (Infections and infestations) | 4 (4) | 7 (7)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (15)
Vomiting (Gastrointestinal disorders) | 7 (7) | 6 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (7)
Insomnia (Psychiatric disorders) | 0 (0) | 6 (7)
Viral upper respiratory tract infection (Infections and infestations) | 5 (5) | 5 (9)
Chronic sinusitis (Infections and infestations) | 1 (3) | 5 (7)
Gastroenteritis (Infections and infestations) | 1 (1) | 5 (5)
Oedema peripheral (General disorders) | 0 (0) | 5 (5)
Pyrexia (General disorders) | 4 (5) | 4 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 4 (6)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 4 (5)
Pharyngitis (Infections and infestations) | 1 (1) | 4 (7)
Migraine (Nervous system disorders) | 1 (4) | 4 (6)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 4 (9)
Infusion site pruritus (General disorders) | 0 (0) | 4 (8)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5)
Somnolence (Nervous system disorders) | 4 (9) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxalta's agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or ≤15 months after study completion. Baxalta requires a review of results communications (eg, for confidential information) ≥30 days prior to submission or communication. Baxalta may request an additional delay of ≤60 days eg, for intellectual property protection.